CLINICAL TRIAL: NCT02579655
Title: Assessing Outcomes of Enhanced Chronic Disease Care Through Patient Education and a Value-based Formulary Study
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Innovates Health Solutions (Other)
Responsible Party: Principal Investigator, Braden Manns, Svare Professor, Health Economics, University of Calgary
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: REB13-1241
Record Dates: First submitted 2015-08-27; First posted 2015-10-19 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Coronary Disease; Stroke; Chronic Kidney Disease; Heart Failure; Diabetes Mellitus; Hypertension; Hypercholesterolemia
MeSH Terms: conditions — Coronary Disease; Stroke; Renal Insufficiency, Chronic; Heart Failure; Diabetes Mellitus; Hypertension; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Copayment Elimination and Personalized Education (Active Comparator): In this arm, participants would have copayment elimination (no cost for preventative medications for hypertension, diabetes, and cardiovascular disease) and free enrollment in a new personalized education program to help participants manage their chronic conditions
  Interventions: Behavioral: Copayment Elimination; Behavioral: Personalized Education
- Copayment Elimination Only (Active Comparator): In this arm, participant's would be randomized to Copayment Elimination (no cost for preventative medications for hypertension, diabetes, and cardiovascular disease) and receive some basic educational information about their chronic disease
  Interventions: Behavioral: Copayment Elimination
- Personalized Education Only (Active Comparator): In this arm, participants would be randomized to free enrollment in a new personalized education program to help patients manage their chronic conditions
  Interventions: Behavioral: Personalized Education
- No intervention (No Intervention): In this arm, participants will have access to some basic online educational information about their chronic disease. There is no intervention in this arm. The comparative group.

INTERVENTIONS:
Behavioral: Copayment Elimination — Patients will receive preventive medications for their chronic conditions free of charge (without the 30% copayment seniors normally pay for their medications)
  Arms: Copayment Elimination Only; Copayment Elimination and Personalized Education
Behavioral: Personalized Education — Tailored Education focusing on optimizing use and adherence to guideline recommended medications, as well as appropriate lifestyle
  Arms: Copayment Elimination and Personalized Education; Personalized Education Only

SUMMARY:
The purpose of this study is to determine the effect of two novel interventions; (1) a value-based formulary which eliminates copayment for selected high-value medications (proven to prevent heart attacks, stroke, and hospitalizations); and (2) a comprehensive patient education program aimed at lifestyle modification and optimal drug use, combined with relay of information on medication use, on the risk of adverse clinical outcomes (mortality, heart attack, stroke, need for coronary revascularization, and chronic disease related hospitalizations) in low-income seniors with chronic conditions over three years of follow-up or until March 31, 2021 (whichever comes first).

DETAILED DESCRIPTION:
Chronic diseases, such as stroke, myocardial infarction, hypertension, diabetes and chronic kidney disease, are the major challenge facing health care systems worldwide. Although medications and lifestyle changes can improve the health of these patients, many do not benefit from these treatments due to barriers at the level of the patient, provider and/or health system, resulting in a care gap. Multiple barriers may contribute to the observed care gap for patients with these chronic diseases-but prior research has identified that 1) out-of-pocket costs for medications (including co-payments); and 2) lack of patient knowledge about the potential benefits of treatment are particularly important. Although these barriers clearly compromise outcomes among people with chronic diseases, the best way to overcome them and close the care gap is uncertain.

In the ACCESS trial, the investigators will study the effect of two novel interventions in 4764 participants with chronic disease. The investigators hypothesize that (1) eliminating copayments for high value cardioprotective medications and (2) a comprehensive patient education program on optimal medication use, combined with relay of information on optimal medication use by the patient to their health care provider, will decrease the risk of adverse clinical outcomes during the follow-up period.

Methods and study design: Parallel, open label, factorial randomized controlled trial with blinded endpoint evaluation assessing the impact of two interventions: 1) elimination of patient copayment for selected medications, and 2) patient education with relay of information to the participant's health care provider.

ELIGIBILITY:
Inclusion Criteria:

>65 years of age (have drug insurance from Alberta Blue Cross with 30% copayment)

Have any one of the following:

* coronary disease
* prior stroke
* chronic kidney disease
* heart failure

OR any two of the following:

* current cigarette smoking (>1/2 pack per day)
* diabetes mellitus
* hypertension
* hypercholesterolemia

Have total family income <$50,000

Exclusion Criteria:

* Coverage by another insurance plan where no drug payment is required (i.e. copayment <30%)
* Inability to participate in education modules (e.g. lack of proficiency in English; cognitive impairment).
* Has every dose of their medication provided to them by a nurse or other professional caregiver?
* Inability to provide informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4764 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Composite rate of all-cause mortality, nonfatal myocardial infarction, nonfatal stroke, need for coronary revascularization, hospitalizations for chronic disease-related ambulatory care sensitive conditions | 3 years or until March 31, 2021 (for patients enrolled after March 31, 2018)
  See below for definitions of individual components for this composite outcome.

SECONDARY OUTCOMES:
All-cause mortality | 3 years or until March 31, 2021 (for patients enrolled after March 31, 2018)
  Die (y/n)
Non-fatal myocardial infarction | 3 years or until March 31, 2021 (for patients enrolled after March 31, 2018)
  Nonfatal MI based on administrative data (y/n)
Non-fatal stroke | 3 years or until March 31, 2021 (for patients enrolled after March 31, 2018)
  Nonfatal stroke based on administrative data (y/n)
Need for coronary revascularization | 3 years or until March 31, 2021 (for patients enrolled after March 31, 2018)
  Coronary revascularization (angioplasty or bypass surgery) based on administrative data (y/n)
hospitalizations for chronic disease-related ambulatory care sensitive conditions | 3 years or until March 31, 2021 (for patients enrolled after March 31, 2018)
  hospitalizations for chronic disease-related ambulatory care sensitive conditions based on administrative data (y/n)
Full adherence to statins | 3 years or until March 31, 2021 (for patients enrolled after March 31, 2018)
  Full adherence to statins will be measured using the proportion of days covered, which is estimated by the "number of days dispensed" / "number of days between prescription renewals" using Alberta Blue Cross data. Patients that have a dispensed supply of statins to cover at least 80% of observed treatment days will be considered adherent (Y/N)
Overall quality of life as measured by the Euroqol EQ5D-5L index score | 3 years or until March 31, 2021 (for patients enrolled after March 31, 2018)
  Index score ranges from 0 to 1 (full health)
Overall health care costs | 3 years or until March 31, 2021 (for patients enrolled after March 31, 2018)
  All costs (cost of interventions taken from study data, and costs of all health care encounters taken from Alberta Health administrative data using grouper codes) will be combined into Canadian $.

CONTACTS AND LOCATIONS:
Overall Officials: Braden Manns, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manns BJ, Tonelli M, Zhang J, Campbell DJ, Sargious P, Ayyalasomayajula B, Clement F, Johnson JA, Laupacis A, Lewanczuk R, McBrien K, Hemmelgarn BR. Enrolment in primary care networks: impact on outcomes and processes of care for patients with diabetes. CMAJ. 2012 Feb 7;184(2):E144-52. doi: 10.1503/cmaj.110755. Epub 2011 Dec 5. PMID 22143232
- [Background] Campbell DJ, King-Shier K, Hemmelgarn BR, Sanmartin C, Ronksley PE, Weaver RG, Tonelli M, Hennessy D, Manns BJ. Self-reported financial barriers to care among patients with cardiovascular-related chronic conditions. Health Rep. 2014 May;25(5):3-12. PMID 24850391
- [Background] Ronksley PE, Sanmartin C, Campbell DJ, Weaver RG, Allan GM, McBrien KA, Tonelli M, Manns BJ, Hennessy D, Hemmelgarn BR. Perceived barriers to primary care among western Canadians with chronic conditions. Health Rep. 2014 Apr;25(4):3-10. PMID 24744042
- [Background] Mann BS, Barnieh L, Tang K, Campbell DJ, Clement F, Hemmelgarn B, Tonelli M, Lorenzetti D, Manns BJ. Association between drug insurance cost sharing strategies and outcomes in patients with chronic diseases: a systematic review. PLoS One. 2014 Mar 25;9(3):e89168. doi: 10.1371/journal.pone.0089168. eCollection 2014. PMID 24667163
- [Background] Ivers NM, Tricco AC, Taljaard M, Halperin I, Turner L, Moher D, Grimshaw JM. Quality improvement needed in quality improvement randomised trials: systematic review of interventions to improve care in diabetes. BMJ Open. 2013 Apr 9;3(4):e002727. doi: 10.1136/bmjopen-2013-002727. Print 2013. PMID 23576000
- [Background] Leibowitz A, Manning WG, Newhouse JP. The demand for prescription drugs as a function of cost-sharing. Soc Sci Med. 1985;21(10):1063-9. doi: 10.1016/0277-9536(85)90161-3. PMID 3936186
- [Background] Keeler EB, Brook RH, Goldberg GA, Kamberg CJ, Newhouse JP. How free care reduced hypertension in the health insurance experiment. JAMA. 1985 Oct 11;254(14):1926-31. PMID 4046121
- [Background] Tamblyn R, Laprise R, Hanley JA, Abrahamowicz M, Scott S, Mayo N, Hurley J, Grad R, Latimer E, Perreault R, McLeod P, Huang A, Larochelle P, Mallet L. Adverse events associated with prescription drug cost-sharing among poor and elderly persons. JAMA. 2001 Jan 24-31;285(4):421-9. doi: 10.1001/jama.285.4.421. PMID 11242426
- [Background] Psaty BM, Lumley T, Furberg CD, Schellenbaum G, Pahor M, Alderman MH, Weiss NS. Health outcomes associated with various antihypertensive therapies used as first-line agents: a network meta-analysis. JAMA. 2003 May 21;289(19):2534-44. doi: 10.1001/jama.289.19.2534. PMID 12759325
- [Background] Gaede P, Vedel P, Parving HH, Pedersen O. Intensified multifactorial intervention in patients with type 2 diabetes mellitus and microalbuminuria: the Steno type 2 randomised study. Lancet. 1999 Feb 20;353(9153):617-22. doi: 10.1016/S0140-6736(98)07368-1. PMID 10030326
- [Background] Demers V, Melo M, Jackevicius C, Cox J, Kalavrouziotis D, Rinfret S, Humphries KH, Johansen H, Tu JV, Pilote L. Comparison of provincial prescription drug plans and the impact on patients' annual drug expenditures. CMAJ. 2008 Feb 12;178(4):405-9. doi: 10.1503/cmaj.070587. PMID 18268266
- [Background] Daw JR, Morgan SG. Stitching the gaps in the Canadian public drug coverage patchwork?: a review of provincial pharmacare policy changes from 2000 to 2010. Health Policy. 2012 Jan;104(1):19-26. doi: 10.1016/j.healthpol.2011.08.015. Epub 2011 Oct 5. PMID 21978939
- [Derived] Campbell DJT, Mitchell C, Hemmelgarn BR, Tonelli M, Faris P, Zhang J, Tsuyuki RT, Fletcher J, Au F, Klarenbach S, Exner DV, Manns BJ; Interdisciplinary Chronic Disease Collaboration. Eliminating Medication Copayments for Low-Income Older Adults at High Cardiovascular Risk: A Randomized Controlled Trial. Circulation. 2023 May 16;147(20):1505-1514. doi: 10.1161/CIRCULATIONAHA.123.064188. Epub 2023 Mar 5. PMID 36871215
- [Derived] Campbell DJT, Tonelli M, Hemmelgarn BR, Faris P, Zhang J, Au F, Tsuyuki RT, Mitchell C, Pannu R, Campbell T, Ivers N, Fletcher J, Exner DV, Manns BJ; Interdisciplinary Chronic Disease Collaboration. Self-Management Support Using Advertising Principles for Older Adults With Low Income at High Cardiovascular Risk: A Randomized Controlled Trial. Circulation. 2023 May 16;147(20):1492-1504. doi: 10.1161/CIRCULATIONAHA.123.064189. Epub 2023 Mar 5. PMID 36871212
- [Derived] Fletcher JM, Saunders-Smith T, Manns BJ, Tsuyuki R, Hemmelgarn BR, Tonelli M, Campbell DJT. Pharmacist and patient perspectives on recruitment strategies for randomized controlled trials: a qualitative analysis. BMC Med Res Methodol. 2020 Oct 31;20(1):270. doi: 10.1186/s12874-020-01140-6. PMID 33129278
- [Derived] Kakumanu S, Manns BJ, Tran S, Saunders-Smith T, Hemmelgarn BR, Tonelli M, Tsuyuki R, Ivers N, Southern D, Bakal J, Campbell DJT. Cost analysis and efficacy of recruitment strategies used in a large pragmatic community-based clinical trial targeting low-income seniors: a comparative descriptive analysis. Trials. 2019 Oct 7;20(1):577. doi: 10.1186/s13063-019-3652-5. PMID 31590686
- [Derived] Campbell DJ, Tonelli M, Hemmelgarn B, Mitchell C, Tsuyuki R, Ivers N, Campbell T, Pannu R, Verkerke E, Klarenbach S, King-Shier K, Faris P, Exner D, Chaubey V, Manns B; Interdisciplinary Chronic Disease Collaboration. Assessing outcomes of enhanced chronic disease care through patient education and a value-based formulary study (ACCESS)-study protocol for a 2x2 factorial randomized trial. Implement Sci. 2016 Sep 26;11(1):131. doi: 10.1186/s13012-016-0491-6. PMID 27671037

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Main analysis SAP (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT02579655/Prot_SAP_001.pdf
  • Statistical Analysis Plan: Secondary analysis SAP - Medication adherence (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT02579655/SAP_002.pdf